CLINICAL TRIAL: NCT02887300
Title: Feasibility Pilot Study to Examine the Role of Mantra Meditation at Reducing Burn Out and Emotional Exhaustion in Emergency Department Staff
Brief Title: Mantra Meditation to Reduce Emotional Exhaustion in Emergency Department Staff
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: Royal College of Physicians (Other); University of Dublin, Trinity College (Other); Health Service Executive, Ireland (Other)
Responsible Party: Principal Investigator, Padraic Dunne, Senior Research Fellow, St. James's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: StJamesH; RCPI (Other: Royal College of Physicians in Ireland); TCD (Other: Trinity College Dublin); HSE (Other: Health Service Executive of Ireland)
Record Dates: First submitted 2016-08-24; First posted 2016-09-02 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Psychological Stress
Keywords: Quality of Health Care; Psychological Stress; Burnout; Health Care Professional; Mantra Meditation; Health Care Economics
MeSH Terms: conditions — Stress, Psychological; Burnout, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive control group (No Intervention): After randomisation, 30 consenting, eligible study participants will be allotted a place in the passive, parallel control group. Participants will work as usual in the ED. Biological and survey samples will be obtained from both groups of participants on the same days:
  T1 - one week before session one T2 - one week after session 4 T3 - three months following T2
- Planned intervention - mantra meditation (Experimental): After randomisation, 30 randomly chosen, ED staff members will be taught mantra meditation by an experienced meditator. Each 4 hour session will occur once every two weeks for 8 weeks (total of 4 sessions) and consist of guided meditation as well as discussions around prescribed texts on the meaning of health care.
  In addition, participants will be asked to engage in home work (20 minutes of a guided mantra meditation on a twice daily basis). Biological and survey samples will be obtained from both groups of participants on the same days:
  T1 - one week before session one T2 - one week after session 4 T3 - three months following T2
  Interventions: Behavioral: Mantra Meditation

INTERVENTIONS:
Behavioral: Mantra Meditation — Week 1:
  20 minute meditation session. Prescribed text discussion. Encouraging a daily practice; the log, daily readings, timer etc.
  Week 2:
  Review of the practice followed by a 20 minute meditation period. Challenges to learning meditation. Second 20 minute meditation. Discussion of prescribed text.
  Week 3:
  20 minute meditation. Review of Atul Gawande's lecture. Second 20 minute period of meditation. Discussion of prescribed text.
  Week 4:
  20 minute meditation session. Discussion of prescribed text. A second 20 minute meditation. End of programme review.
  Arms: Planned intervention - mantra meditation

SUMMARY:
Work in a healthcare setting, such as in an emergency department (ED), while rewarding, can be harmful to psychological well being, as demonstrated by the high numbers of Irish hospital doctors experiencing burnout. Burnout has been linked to poor healthcare quality, medical errors and low patient satisfaction. To prevent further escalation of this problem, there is a need for effective stress-reducing intervention, such as meditation. Meditation practice has a confirmed positive effect on well being; through greater insight and awareness, meditation could help ED staff to become more attentive to and understanding of their patients' complaints, enhancing patient satisfaction and safety. However, based on current research it is difficult to distinguish between the effects of meditation on well being and those associated with bringing people together. There is therefore a need for a larger randomised study (RCT) including a participants that receive no meditation intervention.

This pilot study aims to examine the suitability of RCT to assess the effect of mantra meditation on burnout among ED staff. The investigators will also examine participant recruitment and retention, data management and outcomes assessment methods for well being, patient satisfaction and biological markers. There will be two groups: intervention group (meditation) and control group (non-meditation). 30 ED staff placed in the intervention group will discuss prescribed texts and learn mantra meditation over a 7-week period, accompanied by 20 minutes of daily meditation practice. 30 ED staff placed in the control group will work in the ED as usual and not receive any texts. Biological samples and questionnaires will be obtained at three time points. Participant feedback will also be sought through interviews. This study will highlight issues related to participant recruitment, retention, and adherence, questionnaires, logistics, and data management and pave the way for an efficient, effective, and larger study that will investigate mantra meditation as a means of reducing burnout in ED staff.

DETAILED DESCRIPTION:
The practice of medicine by health care professionals (HCPs), while often meaningful and rewarding, can have a detrimental effect on mental and physical well-being. Alongside the impact of exposure to environmental hazards, doctors are at above-average risk of developing stress-related psychological morbidities, substance abuse, and dysfunctional interpersonal relationships. In particular, the profession of emergency medicine, with its proclivity for complex caseloads, high personal responsibility, and a high-stress environment, can be emotionally and physically arduous. This is corroborated by findings from a recent report by the Royal College of Physicians of Ireland (RCPI), which asserts that high percentage of Irish hospital doctors experience increased levels of burnout. Burnout comprises emotional exhaustion, a diminished sense of personal accomplishment, and depersonalisation, which can manifest as cynicism and a lack of empathy. In light of this, burnout among HCPs can have significant implications for the quality of healthcare provided to patients. Indeed, research demonstrates an association between HCP burnout and reduced compassion and empathy, increased medical errors, and decreased patient satisfaction. There is growing evidence indicating the psychological and physiological benefits of mindfulness and meditation in the general population. While less attention has been afforded to the potential gains for physicians and other HCPs, a limited body of research demonstrates the efficacy of mindfulness-based interventions in improving psychological well being and job satisfaction among this population. For example, a recent pilot study conducted by RCPI demonstrates that mantra meditation significantly reduced emotional exhaustion in 19 HCPs. The enhanced insight and awareness gleaned from meditation can translate into considerable gains for HCPs, patients, and the health service. Meditation can enable HCPs to recognise their own limitations and errors, to listen more attentively, and to observe and understand both physiological and behavioural factors at play. This is corroborated by Beach et al. (Annals of Family Medicine. 2013;11(5):421-8), who found that patients were more likely to give high ratings on clinical communication and to report increased overall satisfaction with clinicians who engage in regular mindfulness practices. Encounters with such clinicians were more likely to be characterised by a patient-centred pattern of communication and conversation about psycho-social issues, while there was no association between clinician mindfulness and discussion of biomedical issues. Meditation also has the potential to enhance patient safety, however, a complex and high-risk system such as healthcare requires additional approaches to augmenting safety. Central to situational awareness, in the context of the health system, is the concept of a mindful clinician who is present in the moment and unencumbered by distraction. In recent years, a state of crisis within Irish healthcare developed, with an increase in the migration of doctors, low levels of recruitment, and under-resourced services. Accordingly, Irish healthcare is characterised by the second-highest level of physician emigration in the world and one of the lowest ratios of doctor/per capita in Europe (www.oecd.org/health/health-at-a-glance-19991312.htm). Reasons for the difficulty in retaining qualified Irish doctors include more favourable working conditions and greater career opportunities abroad. Moreover, the quality of healthcare in Ireland is likely to be compromised by long-term absenteeism if HCPs are forced to leave their jobs prematurely. In light of the unprecedented difficulties in Irish healthcare, and considering the association between HCP burnout and increased absenteeism and disability, the pertinence of this research becomes apparent. HCPs are a vital resource for society and their loss as a result of avoidable ill-health is not only damaging to the health service, but a loss to patients and colleagues. Thus, interventions that aim to reduce or prevent burnout and stress-related psychological morbidities in HCPs are urgently required.

ELIGIBILITY:
Inclusion Criteria:

* Staff member (nurse or doctor) of the ED department of St. James' hospital, Dublin
* Preference to participate in the study

Strict inclusion criteria will be applied for admitted ED patients (determined by the Clinical Research Facility data controller and ward staff):

* Conscious patient
* Cognitively functioning to an adequate level
* Not actively abusing any substance
* Preference to participate
* Over the age of 18 years

Exclusion Criteria:

* Alcohol or substance abuse within the past 6 months
* Are currently using (at the time of enrolment) anti-psychotic medication or recently started on anti-depressant medication (less than 3 months at the time of enrolment). Participants on a stable dose of anti-depressant medication (for more than 3 months) will be permitted but advised to consult with their GP or psychiatrist prior to enrolment.
* A diagnosis of schizophrenia
* More than 4 consecutive classes of meditation training or mind-body practices (including yoga and tai-chi) in the past 2 years
* Current pregnancy or lactation
* Not available to attend all programme dates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-06-23 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ED staff burn out using the Maslach Burnout Inventory (MBI) | Week 8 and 20

SECONDARY OUTCOMES:
Change from baseline in retention and adherence of consenting participants to both arms of the study | Week 8 and 20
Change from baseline in ED staff anxiety and depression using the Depression, Anxiety and Stress Scale (DASS) | Week 8 and 20
Change from baseline in ED staff response to meditation using the Five Facets Mindfulness Scale (FFMS) at week 8 and 20 | Week 8 and 20
Change from baseline in ED staff professional quality of life using the Professional Quality of Life Scale (PQoLS) | Week 8 and 20
Change from baseline in participant 24 h ambulatory blood pressure | Week 8
Change from baseline in participant heart rate using Fitbit device | Week 8
Change from baseline in participant salivary cortisol using ELISA on week 8 | Week 8
Number of participants in the intervention group adhering to home meditation practice using a bespoke application linked to a Fitbit device. | Week 8
Participant feedback on intervention through qualitative structured interviews | Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Barry White, MD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Trinity Health Centre, Centre for Learning and development, SJH, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Patient identity will be coded by a designated data controller from the Wellcome/Health Research Board Clinical Research Facility, St James' Hospital. Therefore, only individual participant data in the form of coded data will be shared via academic publications only.

REFERENCES:
- [Background] Hayes B, Fitzgerald D, Doherty S, Walsh G. Quality care, public perception and quick-fix service management: a Delphi study on stressors of hospital doctors in Ireland. BMJ Open. 2015 Dec 23;5(12):e009564. doi: 10.1136/bmjopen-2015-009564. PMID 26700286
- [Background] Prinz P, Hertrich K, Hirschfelder U, de Zwaan M. Burnout, depression and depersonalisation--psychological factors and coping strategies in dental and medical students. GMS Z Med Ausbild. 2012;29(1):Doc10. doi: 10.3205/zma000780. Epub 2012 Feb 15. PMID 22403595
- [Background] Amtul Z, Arena A, Hirjee H, Khan ZU, Maldeniya PM, Newman RI, Burhan AM, Wetmore S, Vasudev A. A randomized controlled longitudinal naturalistic trial testing the effects of automatic self transcending meditation on heart rate variability in late life depression: study protocol. BMC Complement Altern Med. 2014 Aug 19;14:307. doi: 10.1186/1472-6882-14-307. PMID 25134497
- [Background] Beach MC, Roter D, Korthuis PT, Epstein RM, Sharp V, Ratanawongsa N, Cohn J, Eggly S, Sankar A, Moore RD, Saha S. A multicenter study of physician mindfulness and health care quality. Ann Fam Med. 2013 Sep-Oct;11(5):421-8. doi: 10.1370/afm.1507. PMID 24019273
- [Background] Nieuwenhuijsen K, de Boer AG, Verbeek JH, Blonk RW, van Dijk FJ. The Depression Anxiety Stress Scales (DASS): detecting anxiety disorder and depression in employees absent from work because of mental health problems. Occup Environ Med. 2003 Jun;60 Suppl 1(Suppl 1):i77-82. doi: 10.1136/oem.60.suppl_1.i77. PMID 12782751
- [Background] Carlson LE, Speca M, Faris P, Patel KD. One year pre-post intervention follow-up of psychological, immune, endocrine and blood pressure outcomes of mindfulness-based stress reduction (MBSR) in breast and prostate cancer outpatients. Brain Behav Immun. 2007 Nov;21(8):1038-49. doi: 10.1016/j.bbi.2007.04.002. Epub 2007 May 22. PMID 17521871
- [Background] Ryan M, Gerard K. Using discrete choice experiments to value health care programmes: current practice and future research reflections. Appl Health Econ Health Policy. 2003;2(1):55-64. PMID 14619274
- [Derived] Dunne PJ, Lynch J, Prihodova L, O'Leary C, Ghoreyshi A, Basdeo SA, Cox DJ, Breen R, Sheikhi A, Carroll A, Walsh C, McMahon G, White B. Burnout in the emergency department: Randomized controlled trial of an attention-based training program. J Integr Med. 2019 May;17(3):173-180. doi: 10.1016/j.joim.2019.03.009. Epub 2019 Mar 29. PMID 30956141